CLINICAL TRIAL: NCT02580357
Title: Comparison of Two Different Low-level Laser Intensity Protocols on the Healing of Palatal Wounds After Connective Tissue Graft Removal: Randomized Clinical Trial
Brief Title: Comparison of Two Different Low-level Laser Intensity Protocols on the Healing of Palatal Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UEPJMF 2
Record Dates: First submitted 2015-10-09; First posted 2015-10-20 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-03

CONDITIONS: Palatal Wound
Keywords: Connective tissue graft; Gingival recession; Low level laser therapy
MeSH Terms: conditions — Gingival Recession | interventions — Low-Level Light Therapy; Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Level Laser therapy (LLLT) Sham (Sham Comparator): The patients allocated to the control group received sham irradiation. For this, black rubber protection was placed at the tip of the laser device, which did not allow the light to reach the tissue. The applications were performed by a different operator (CAS) from the one who measured the study parameters. During irradiation, the tip of the laser probe was placed perpendicularly with slight contact on the area. Laser therapy was initiated in the immediate postoperative period (just after sutures) and was repeated by six more applications performed every other day, with a total of 7 laser applications.
  Interventions: Procedure: Low Level Laser Therapy; Device: GaAlAs laser
- GaAlAs Laser therapy (LLLT) 60 J/cm² (Experimental): The irradiation was performed with a GaAlAs diode laser that continuously emitted a wavelength of 660 nm with a power of 30 mW. The patients allocated for the group 60 received the following protocol for laser application: Two (2) points of irradiation were performed using a total energy density (fluence) of 60 J/cm2 and a time of 60 seconds (30 J/cm2 per point and an application time of 30 seconds per point). During irradiation, the tip of the laser probe was placed perpendicularly with slight contact on the area. Laser therapy was initiated in the immediate postoperative period (just after sutures) and was repeated by six more applications performed every other day, with a total of 7 laser applications. The power of the equipment was calibrated prior to each application.
  Interventions: Procedure: Low Level Laser Therapy; Device: GaAlAs laser
- GaAlAs Laser therapy (LLLT) 30 J/cm² (Experimental): The irradiation was performed with a GaAlAs diode laser that continuously emitted a wavelength of 660 nm with a power of 30 mW. The patients allocated for the group 30 received the following protocol for laser application: Two (2) points of irradiation were performed using a total energy density (fluence) of 30 J/cm2 and a time of 30 seconds (15 J/cm2 per point and an application time of 15 seconds per point). During irradiation, the tip of the laser probe was placed perpendicularly with slight contact on the area. Laser therapy was initiated in the immediate postoperative period (just after sutures) and was repeated by six more applications performed every other day, with a total of 7 laser applications. The power of the equipment was calibrated prior to each application.
  Interventions: Procedure: Low Level Laser Therapy; Device: GaAlAs laser

INTERVENTIONS:
Procedure: Low Level Laser Therapy — Low Level Laser Therapy on the palatal donor site of connective tissue graft.
  Other Names: Laser stimulation
Device: GaAlAs laser — Utilization of GaAlAs laser to irradiation on the palatal donor site.
  Other Names: Low level GaAlAs laser

SUMMARY:
The aim of this study was to compare two intensities of LLLT on wound healing process of the donor palatine area after CTG removal.

DETAILED DESCRIPTION:
This is a prospective, parallel and controlled clinical trial. The population evaluated in the study was selected at Science and Technology Institute - ICT- São José dos Campos, College of Dentistry.

Patients were assigned to one of the three treatment groups:

* Group 60 (Test, n=18): Periodontal surgery for root coverage through connective tissue graft and LLLT application on donor site using a 60 J/cm² dose.
* Group 30 (Test, n=18): Periodontal surgery for root coverage through connective tissue graft and LLLT application on donor site using a 30 J/cm² dose.
* Group Sham (Control, n= 18): Periodontal surgery for root coverage through connective tissue graft and LLLT SHAM on donor site.

All surgeries were performed by the same expert periodontist (MPS). Before the surgical procedure, all patients were enlightened about the causes and consequences of gingival recession and prevention techniques. Factors related to the origin of gingival recession, such as toothbrush trauma and inflammation caused by biofilm, were controlled through instruction on standardized brushing technique to avoid the influence of other hygiene methods capable of promoting trauma on soft tissues. Standardized dental floss and toothbrushes were given to patients. The surgical technique adopted in the recession defects was the trapezoidal-type of CAF and the connective tissue graft was removed from palate mucosa . Briefly, a first incision on the palate was performed perpendicularly to the long axis of the teeth, 2 to 3 mm apical to the gingival margin. The mesial-distal length of the incision was determined by the length of the graft required to cover the recession. Because the selected recessions were in maxillary canines and premolars, the lengths of the graft varied minimally (10-12mm). The second incision was made parallel to the first one (1-2 mm apically and parallel to the long axis of the teeth) to separate the subepithelium connective tissue from the epithelial layer. The incision is carried far enough apically to provide a 7- mm height of connective tissue to cover the denuded root surface. Afterward, another incision parallel to the long axis of the teeth starting from the first incision was performed to separate the subepithelium connective tissue from the periosteum. Then, the connective tissue graft was removed from the palate as atraumatically as possible. Single sutures were made on the palate (4-0 silk) and the graft was sutured on the receptor site.

The evaluated parameters were wound remaining area (WRA), scar and tissue colorimetry (TC), tissue thickness (TT) and postoperative discomfort (D), evaluated at baseline and 7, 14, 45, 60, and 90 days after surgery.

Statistical Analysis: All data were expressed as mean ± standard deviation or expressed in percentages during the descriptive phase. Data were analyzed according to distribution by the Shapiro-Wilk test. For the remaining wound area, tissue colorimetry, tissue thickness, and postoperative discomfort parameter analysis, two way repeated measures ANOVA was performed for intra- and intergroup analysis. T test was used for intergroup comparison of the number of analgesics taken. The presence or absence of scars was measured by Q-square test. Statistical analysis was performed using Sigma Plot 12.0. In all tests a significance level of 0.05 was chosen.

ELIGIBILITY:
Inclusion Criteria:

* Patients were 20 to 70 years old and of both genders, presenting Class I or II Miller gingival recession on vital canines or premolars in the palatine region (donor site) with no pathological or morphological alterations.
* Patients agreed to and signed the formal consent to participate in the study after receiving an explanation of risks and benefits from an individual who was not a member of the present study (Resolution no. 196 - October, 1996, and Ethics and Code of Professional Conduct in Dentistry - CFO 179/93).

Exclusion Criteria:

* Were excluded patients with systemic problems that contraindicated surgical procedure
* Those under medication that could interfere with the wound healing
* Those who smoked
* Those who were pregnant or lactating, and
* Those who had had periodontal surgery on the study area.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-02; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mauro P Santamaria, PhD, Principal Investigator — College of Dentistry - São José dos Campos, State University of São Paulo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zucchelli G, Amore C, Sforza NM, Montebugnoli L, De Sanctis M. Bilaminar techniques for the treatment of recession-type defects. A comparative clinical study. J Clin Periodontol. 2003 Oct;30(10):862-70. doi: 10.1034/j.1600-051x.2003.00397.x. PMID 14710766
- [Background] Bruno JF. Connective tissue graft technique assuring wide root coverage. Int J Periodontics Restorative Dent. 1994 Apr;14(2):126-37. PMID 7928129
- [Derived] da Silva Neves FL, Silveira CA, Dias SB, Santamaria Junior M, de Marco AC, Kerbauy WD, de Melo Filho AB, Jardini MA, Santamaria MP. Comparison of two power densities on the healing of palatal wounds after connective tissue graft removal: randomized clinical trial. Lasers Med Sci. 2016 Sep;31(7):1371-8. doi: 10.1007/s10103-016-1988-6. Epub 2016 Jun 25. PMID 27344670

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At clinical site
Period: Overall Study
Arm/Group | Low Level Laser Therapy (LLLT) Sham | GaAlAs Laser Therapy (LLLT) 60 J/cm² | GaAlAs Laser Therapy (LLLT) 30 J/cm²
Started | 18 | 18 | 18
Completed | 15 | 18 | 18
Not Completed | 3 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Level Laser Therapy (LLLT) Sham | GaAlAs Laser Therapy (LLLT) 60 J/cm² | GaAlAs Laser Therapy (LLLT) 30 J/cm² | Total
Number analyzed (Participants) | 15 | 18 | 18 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 18 | 18 | 51
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.01 (7.6) | 43.2 (9.8) | 47 (9.3) | 43.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 11 | 32
  Male | 7 | 5 | 7 | 19
Region of Enrollment [Number; unit: participants]
  Brazil | 15 | 18 | 18 | 51
Remaining wound area (RWA-mm2 ) [Mean (Standard Deviation); unit: square millimeters] | 62.91 (23.27) | 50.15 (18.49) | 65.74 (25.08) | 59.6 (22.28)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Remaining Wound Area (RWA)
Description: For this, standardized photographs were taken (brightness, distance and angle). A scale was used as a reference to measure this area. These photographs were exported to image software ( Image J - NIH, Bethesda, USA) and remaining wound area was measured in square millimeters (mm²).
Time Frame: 7,14, 45 and 60 post operative days
Measure: Mean (Standard Deviation); unit: Square millimeters
Units Other Than Participants: Photographs
Arm/Group | Low Level Laser Therapy (LLLT) Sham | GaAlAs Laser Therapy (LLLT) 60 J/cm² | GaAlAs Laser Therapy (LLLT) 30 J/cm²
Number analyzed (Participants) | 15 | 18 | 18
Number analyzed (Photographs) | 60 | 72 | 72
Square millimeters
  RWA 7 days | 62.91 (23.27) | 50.15 (18.49) | 65.74 (25.08)
  RWA 14 days | 29.86 (21.84) | 28.38 (13.89) | 27.67 (16.16)
  RWA 45 days | 6.63 (11.85) | 8.17 (6.66) | 7.45 (7.93)
  RWA 60 days | 5.52 (9.37) | 2.33 (2.95) | 3.08 (2.96)

2. Secondary Outcome: Postoperative Discomfort
Description: After air jet application, patients were requested to score postoperative discomfort through on a visual analogue scale (VAS) of 10 centimeters, in which 0 meant "no pain" and 10 meant "extreme pain". After this, a postoperative discomfort average for all groups was obtained.
Time Frame: 7, 14, 45, and 60 days after surgical procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Level Laser Therapy (LLLT) Sham | GaAlAs Laser Therapy (LLLT) 60 J/cm² | GaAlAs Laser Therapy (LLLT) 30 J/cm²
Number analyzed (Participants) | 15 | 18 | 18
units on a scale
  Pain 7 days | 0 (0) | 0 (0) | 0 (0)
  Pain 14 days | 0 (0) | 0 (0) | 0 (0)
  Pain 45 days | 0 (0) | 0 (0) | 0 (0)
  Pain 60 days | 0 (0) | 0.056 (0.23) | 0 (0)

3. Other Pre Specified Outcome: Tissue Thickness
Description: Through four fixed points marked 5 and 7 mm from the gingival margin in the operated region, tissue thickness of palatine masticatory mucosa. One stent was made to standardize the points to be measured. The stent was positioned, and with a periodontal probe and the points were marked. Then the stent was removed and measurements were taken. For this, an endodontic spacer with a rubber cursor was put on the marked points for it to reach the palatine bone plate. Then the cursor was taken to the tissue carefully to not pressuring it. The distance between the spacer tip and the cursor was measured using a digital pachymeter and measured in millimeters (mm).
Time Frame: Before the procedure and 3 months after the procedure
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Low Level Laser Therapy (LLLT) Sham | GaAlAs Laser Therapy (LLLT) 60 J/cm² | GaAlAs Laser Therapy (LLLT) 30 J/cm²
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/15 | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No